CLINICAL TRIAL: NCT05938231
Title: A Prospective, Multicenter, Randomized Controlled Clinical Study to Evaluate the Safety and Performance of the Gastric Bypass Stent System as a Weight Loss Treatment for Obesity
Brief Title: Tangji Gastric Bypass Stent Study for Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Tangji Medical Technology Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HZTG01
Record Dates: First submitted 2023-06-02; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Diet Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- trial group (Experimental): In the trial group, the patients are treated with Gastric Bypass Stent System implanted under the gastroscope as well as the dietary intervention; The trial is carried out for 9 months, of which in the trial group, the patients have 3-month treatment period and then have 6-month follow-up period after the Gastric Bypass Stent System is removed.
  Interventions: Device: Gastric Bypass Stent System; Behavioral: Dietary Intervention
- control group (Other): In the control group, the patients are treated only with dietary intervention; the patients have 9-month dietary intervention in the corresponding period.
  Interventions: Behavioral: Dietary Intervention

INTERVENTIONS:
Device: Gastric Bypass Stent System — Subjects will be treated with the Gastric Bypass Stent System implanted under gastroscopy. Following a 3-month treatment period, the device is removed, and subjects are followed for 6 months.
  Arms: trial group
Behavioral: Dietary Intervention — The patients in the trial group or in the control group,have 9-month dietary intervention in the syudy period.

SUMMARY:
The Gastric Bypass Stent System is intended to be used in weight loss treatment for obesity in patients with a BMI ≥ 30 kg/m2. In this clinical investigation the Sponsor seeks to demonstrate the safety and performance of the Gastric Bypass Stent System for its proposed indication in weight loss treatment for obesity in the China.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-60 years, both male and female;
2. Obese patients with BMI ≥ 30 kg/m2, who are willing to be treated with Gastric Bypass Stent System or dietary intervention;
3. Patients with ASA I~II grade;
4. The patient understands the onjective of the trial and is volunteered to participate in the trial and has signed the Informed Consent Form (ICF).

Exclusion Criteria:

1. Have a weight loss of more than 4.5 kg in the past three months, or take weight-loss drugs in the past month;
2. Patients who used non-steroidal anti-inflammatory drugs (NSAIDs) and corticosteroids in the past month;
3. Patients diagnosed with type 1 diabetes;
4. Patients with the function of islet β cell basically lost, C-peptide ≤ 1/2 of the normal low limit or low and flat C-peptide release curve under glucose load;
5. Patients with iron deficiency or iron deficiency anemia;
6. Patients with coagulation dysfunction who used aspirin and other anticoagulants in the past month;
7. Patients with severe liver and kidney dysfunction, and the serum creatinine concentration of greater than 180 μmol/L;
8. Patients with Class III heart function of NYHA or higher, or pulmonary dysfunction;
9. Patients who have undergone ERCP procedure, or have a history of cholecystitis or liver abscess;
10. Patients with duodenal ulcer, gastric ulcer or previous and existing pancreatitis;
11. Patients with gallstones (diameter ≥ 20 mm) with clinical symptoms;
12. Patients with thyroid dysfunction;
13. Patients with hemorrhage or potential hemorrhage in the digestive tract;
14. Patients with gastrointestinal tract anomalies, such as gastrointestinal tract atresia, or other conditions that would result in failed placement in the gastrointestinal tract;
15. Patients with a history of bowel obstruction or related diseases in the past year;
16. Patients with a history of systemic lupus erythematosus or scleroderma;
17. Patients with severe infections that are not controlled, not suitable for a procedure;
18. Patients with poor general condition and having endoscopic contraindications (as evaluated by the investigator);
19. Pregnant women or women having the plan for pregnancy;
20. Drug abusers or alcohol addicts or patients with uncontrollable mental illness;
21. Patients who participated in other clinical trials of drugs or medical devices before enrollment and do not reach the endpoint time limit;
22. Patients who participated in other clinical trials of drugs or medical devices before enrollment 3 months.
23. Patients with any other conditions evaluated by the investigators as unsuitable for participating in the trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
EWL% at 3 months after device implantation procedure. | 3 months after device implantation procedure
  EWL%=(Preoperative weight - Weight at follow-up)/(Preoperative weight - Body weight at BMI of 25 kg/m2)*100%.

SECONDARY OUTCOMES:
Evaluation of device use in the trial group | Baseline visit V2 and 1, 3 months after the procedure
  Gastroscopy will be performed During the procedure (Visit 2) and at device removal(Visit 5).The user assesses whether the Gastric Bypass Stent can be used successfully during the procedure.
  Abdominal X-ray will be performed 1 month after the implantation procedure (Visit 4) and before Gastric Bypass Stent retrieval (Visit 5). An abdominal plain film will be used to assess the status of the Gastric Bypass Stent.The stent is completely located in the duodenal bulb the stent is unfolded, and the outline is clear.
Difference in BMI change from baseline between the two groups at 1, 3, 4, 6 and 9 months after the patients are enrolled | from baseline to 1, 3, 4, 6, and 9 months after the procedure.
Changes in HbA1c at 3, 6 and 9 months after the patients are enrolled | 3, 6, and 9 months after the procedure
Drug dose of hypoglycemic agents at 1, 3, 4, 6 and 9 months after the patients are enrolled | 1, 3, 4, 6, and 9 months after the procedure
Changes in blood glucose-related indicators of the patients from Baseline | from baseline to 1, 3, 4, 6, and 9 months after the procedure.
  Through observe the changes of (fasting insulin, fasting blood glucose, fasting C-peptide) from baseline to 1, 3, 4, 6, and 9 months to evaluate whether implanting the investigational device will bring any changes to patients' blood glucose.
Difference in blood lipid change from baseline (TC, TG, HDL-C, LDL-C) at 3, 4, 6, and 9 months after the patients are enrolled | from baseline to 3, 4, 6, and 9 months after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Shutian Zhang, Principal Investigator — Beijing Friendship Hospital
Locations (7):
- China (7):
  - Beijing Friendship Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Beijing Shijitan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Nanjing Drum Tower hospital, Nanjing, Jiangsu
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The Affiliated Hospital of lnner Mongolia Medical University, Hohhot, Neimenggu
  - Tangdu Hospital,Fouth Military Medical University, Xi’an, Shanxi
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No